CLINICAL TRIAL: NCT00385034
Title: Computer-assisted Screening for Intimate Partner Violence in Family Practice - a Randomized Controlled Trial
Brief Title: Computer-assisted Screening for Intimate Partner Violence in Family Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AL-777601096-01; CIHR Fellowship: 17744; CIHR/OWHC Fellowship: 24050
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Screening for Partner Violence
Keywords: randomized controlled trial; RCT; partner violence; IPV; screening; family practice; computer

INTERVENTIONS:
Device: Interactive computer based health-risk survey before doctor's visit

SUMMARY:
This study tested the effectiveness of computer-assisted screening for identifying patients at risk of intimate partner violence (IPV) in a Canadian family practice. It was hypothesized that the use of computer-assisted screening among female patients would lead to higher rates of IPV discussion-opportunity and IPV detection during medical consultations, compared to patients receiving standard medical care.

ELIGIBILITY:
Inclusion Criteria:

* woman
* at least 18 years of age
* visiting one of the participant physicians
* in a current or recent intimate relationship during the last 12 months
* having the ability to speak and read English and give consent

Exclusion Criteria:

* visiting a provider other than the regular family physician
* new patient
* previously approached for the study
* very sick
* had a dual appointment (herself and accompanied dependent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2005-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Discussion-opportunity about risk of partner abuse during physician-patient medical encounter (audiotaped data)
Detection of partner abuse during physician-patient medical encounter (audio taped data)

SECONDARY OUTCOMES:
Patient acceptance of the computer-assisted screening(paper-pencil exit survey)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Levinson, MD, FRCPC, Principal Investigator — St. Michael's Hospital and University of Toronto; Farah Ahmad, PhD(student), Principal Investigator — St. Michael's Hospital and University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ahmad F, Skinner HA, Stewart DE, Levinson W. Perspectives of family physicians on computer-assisted health-risk assessments. J Med Internet Res. 2010 May 7;12(2):e12. doi: 10.2196/jmir.1260. PMID 20457555
- [Derived] Ahmad F, Hogg-Johnson S, Stewart DE, Skinner HA, Glazier RH, Levinson W. Computer-assisted screening for intimate partner violence and control: a randomized trial. Ann Intern Med. 2009 Jul 21;151(2):93-102. doi: 10.7326/0003-4819-151-2-200907210-00124. Epub 2009 Jun 1. PMID 19487706